CLINICAL TRIAL: NCT06812715
Title: Clonal Dynamics of Chronic Lymphocytic Leukaemia Treated With Pirtobrutinib After Previous Treatment With Zanubrutinib
Acronym: PIPOZA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/028
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Pirtobrutinib; Bruton Tyrosine Kinase; BTK mutation; clonal dynamics; CLL; BTK inhibitor; Chronic Lymphocytic Leukaemia; Leukaemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Leukemia | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): In this single-arm study, patients will receive 200mg of pirtobrutinib once daily on Day 1-28 of each 28-day cycle.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Pirtobrutinib is a first-in-class, oral noncovalent Bruton tyrosine kinase (BTK) inhibitor (BTKi) that was approved in January 2023 in the United States for the treatment of relapsed/refractory (R/R) mantle cell lymphoma (MCL) and later that same year CLL. It is currently being investigated across several global randomised phase III trials for frontline and R/R chronic lymphocytic leukaemia (CLL).

SUMMARY:
This is a multicentre single-arm prospective phase II trial evaluating pirtobrutinib in the treatment of relapsed/refractory (R/R) Chronic Lymphocytic Leukaemia (CLL) patients who have previously received zanubrutinib, and to specifically evaluate Bruton Tyrosine Kinase (BTK) mutational status (clonal dynamics) before, during and after treatment with pirtobrutinib.

DETAILED DESCRIPTION:
Following confirmation of eligibility and registration to the study, patients will receive treatment with pirtobrutinib until progressive disease (PD) according to International Workshop on Chronic Lymphocytic Leukaemia (iwCLL) 2018 criteria, unacceptable toxicity, or patient withdrawal. Following first progression, treatment may continue if in the opinion of the investigator the patient is deriving clinical benefit.

BTK mutational status and analysis of CLL clonal dynamics on peripheral blood will be performed prior to the first dose of treatment, Day 1 of each cycle thereafter while on study treatment, End of Treatment (EoT), and at time of PD.

Response will be assessed by the investigator based on physical examination, CT scan (or MRI), haematology results, and bone marrow examinations according to iwCLL 2018 response criteria.

Patients who discontinue treatment for any reason will have an EoT visit within 7 days after the last dose of treatment or decision to cease treatment. Additionally, they will have a Safety Follow-up visit 28 days + 7 days after the last dose of treatment or decision to discontinue treatment. Following these two visits, patients will move into the Follow-up Phase of the study where they will be assessed every 12 weeks ± 4 weeks. Patients with PD will be followed for survival and new anti-CLL therapy only. All patients will be followed up until the last registered patient has been on pirtobrutinib for 36 months without PD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent using the PIPOZA Patient Information and Consent Form (PICF)
2. Confirmed diagnosis of CLL according to iwCLL 2018 criteria, also including CLL with atypical immunophenotype
3. Prior systemic therapy, which must include zanubrutinib as the most recent prior line of therapy. Patients must have received at least one cycle (28 days) of zanubrutinib
4. Patients must have an indication for second- or subsequent-line treatment in the opinion of the investigator as defined by iwCLL 2018 criteria, including:

   * Where the original indication for treatment has not resolved with initial therapy and it is considered reasonable to initiate second-line treatment without waiting for formal disease progression to be manifest
   * Where the rate of disease progression is considered rapid, and initiation of subsequent therapy is considered acceptable before formal progression where there is substantial persisting disease burden
5. Age 18 years of age or older at time of signing the PICF
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
7. Must have adequate bone marrow function, as defined below:

   * Absolute neutrophil count > 0.75 × 109/L; if marrow is known to be infiltrated by CLL, granulocyte-colony stimulating factor (G-CSF) support may be used to achieve eligibility criteria
   * Platelets ≥ 30 × 109/L independent of transfusions within 7 days prior to screening assessment
   * Haemoglobin ≥ 70 g/L independent of transfusions within 7 days prior to screening assessment
8. Normal hepatic function defined as:

   * Total bilirubin ≤ 1.5× upper limit of normal (ULN) or ≤ 3.0 x ULN with documented liver involvement and/or Gilbert's Disease
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 × ULN or ≤ 5.0 × ULN with documented liver involvement
9. Adequate renal function defined as creatinine clearance of > 30 mL/minute calculated by Cockroft-Gault formula or using biochemical or nuclear medicine techniques
10. Ability to swallow tablets
11. Patients must have had a zanubrutinib washout period of at least 24 hours prior to the planned start date of pirtobrutinib on Day 1 Cycle 1
12. Prior treatment-related adverse events must have recovered to Grade ≤ 1 or pretreatment baseline with the exception of alopecia and Grade 2 peripheral neuropathy
13. Women of childbearing potential defined as not postmenopausal for at least 2 years or surgically sterile must have a negative serum pregnancy test documented within 14 days prior to planned started date of pirtobrutinib on Day 1 Cycle 1
14. Men with partners of childbearing potential or women of childbearing potential must agree to use a highly effective contraceptive method of birth control during study treatment and for at least 6 months following the last dose of study drug. Sperm donation is prohibited during the duration of participation in this study and for 6 months after the last dose of study drug. Acceptable methods of birth control are:

    * Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally
    * Progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant
    * Intrauterine device Intrauterine hormone-releasing system
    * Bilateral tubal occlusion
    * Vasectomised partner
    * Sexual abstinence: Considered a highly effective method only if defined as refraining from heterosexual intercourse during an entire period of risk associated with the study treatment. The reliability of sexual abstinence needs will be evaluated in relation to the duration of the study and to the usual lifestyle of the patient
15. The patient understands the purpose of the trial and procedures required for the trial which includes compliance with the protocol requirements and restrictions listed in the PICF and in this protocol

Exclusion Criteria:

1. Known or suspected Richter's Transformation to diffuse large B-cell lymphoma, prolymphocytic leukaemia, or Hodgkin lymphoma at any time prior to registration
2. Known or suspected history of central nervous system involvement
3. History of allogeneic or autologous stem cell transplant or chimeric antigen receptor T-cell (CAR-T) therapy within the past 60 days and/or with any of the following:

   * Active graft versus host disease
   * Cytopenias from incomplete blood cell count recovery post-transplant or CAR-T therapy
   * Need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity Grade > 1 from CAR-T therapy
   * Ongoing immunosuppressive therapy
4. Positive serology for human immunodeficiency virus (HIV) test in Screening 5. Concurrent anticancer therapy

6. Use of ≥ 20 mg prednisone QD or equivalent dose of steroid per day within 7 days prior to the planned pirtobrutinib start date on Day 1 Cycle 1. Patients may not be on prednisone of any dose intended for antineoplastic use 7. Vaccination with a live vaccine within 28 days prior to registration 8. Prolongation of the corrected QT interval using the Fredericia formula (QTcF) > 470 msec (QTcF is calculated using Fridericia's Formula: QTcF = QT / [RR0.33])

* Correction of suspected drug induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation
* Manual correction for underlying bundle branch block is allowed Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker 9. Female patient who is pregnant or plans to become pregnant within 1 month after the last dose of study treatment 10. Female patient who is lactating or plans to breastfeed during the study or within 1 week after the last dose of study drug 11. Active second malignancy 12. Clinically significant active malabsorption syndrome including surgical resection of small intestine or other condition likely to affect gastrointestinal (GI) absorption of the oral administered study drugs 13. Active hepatitis B or C infection defined as:
* Hepatitis B virus (HBV): positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (anti-HBc). If anti-HBc positive with surface antigen negative, patient will need to have a negative result for hepatitis B DNA before start of study therapy. Patients who are anti-HBc positive and hepatitis B polymerase chain reaction positive will be excluded
* Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before start of study therapy. Patients who are hepatitis C RNA positive will be excluded 14. Known active cytomegalovirus infection Note: Patients with an unknown or negative status are eligible 15. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, parasitic, or fungal) or other clinically significant active disease process which, in the opinion of the investigator, may pose a risk for patient participation. Screening for chronic conditions is not required 16. Active uncontrolled auto-immune cytopenia (e.g., autoimmune haemolytic anaemia, idiopathic thrombocytopenic purpura) where new therapy is introduced, or concomitant medication escalated within the 4 weeks prior to registration is required to maintain adequate blood counts. Stable controlled auto-immune cytopenias are allowed as long as required blood count criteria are met 17. Prior treatment with pirtobrutinib 18. Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist 19. Known hypersensitivity to any component or excipient of pirtobrutinib 20. Significant cardiovascular disease defined as:
* Unstable angina or acute coronary syndrome within the past 2 months prior to registration
* History of myocardial infarction within 3 months prior to registration
* Documented left ventricular ejection fraction by any method of ≤ 40% in the 12 months prior to registration
* ≥ Grade 3 New York Heart Association functional classification system of heart failure
* Uncontrolled or symptomatic arrhythmias 21. History of uncontrolled or symptomatic arrhythmias including Grade ≥ 3 arrhythmia on a prior BTKi 22. History of major bleeding on a prior BTKi NOTE: Major bleeding is defined as bleeding having 1 or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the Hb level of at least 20 g/L; or bleeding in a critical area or organ (e.g., retroperitoneal, intra-articular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome) 23. History of stroke or intracranial haemorrhage within 6 months prior to registration 24. Major surgery within 4 weeks prior to registration 25. History of bleeding diathesis 26. Current treatment with strong P-glycoprotein (P-gp) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Cloncal dynamics of BTK mutations in CLL before, during and after treatment with pirtobrutinib | Before the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease

SECONDARY OUTCOMES:
Overall response rate in CLL with pirtobrutinib after prior immediate zanubrutinib | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
The efficacy as assessed by time to response (TTR) | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The time from the start of pirtobrutinib to the first objective response observed for patients who achieves a complete remission (CR), complete remission with an incomplete marrow recovery (CRi), nodular partial remission (nPR), partial remission (PR) or the initiation of subsequent anticancer therapy. TTR also includes partial remission with lymphocytosis (PR-L) as sensitivity analysis
Efficacy as assessed by Duration of Response (DOR) | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The time from onset of a CR, CRi, nPR, PR to the earlier of the documentation of definitive progressive disease ([PD] per iwCLL 2018 criteria) or death from any cause, whichever occurred first. Duration of response and time to response will be evaluated for responders (CR, CRi, nPR, PR) only. DOR including PR-L as a response will be analysed with the same method as DOR
Efficacy as assessed by Disease Control Rate (DCR) | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The percentage of patients who have achieve CR, CRi, nPR, PR, PR-L, or SD
Efficacy as assessed by Time to next treatment (TTNT) | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The time from the date of first pirtobrutinib dose (Day 1 Cycle 1) to the date of the initiation of the next systemic anticancer therapy for CLL or death from any cause, whichever occurs first
Efficacy as assessed by progression free survival | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The time from the date of first pirtobrutinib dose (Cycle 1 Day 1) until PD (per iwCLL 2018 criteria) or death from any cause, whichever occurs first
Efficacy as assessed by overall survival | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  The time from first pirtobrutinib dose (Day 1 Cycle 1) until death from any cause. If the patient is alive or lost to follow-up at the time of data analysis, OS data will be censored on the last date the patient is known to be alive
Adverse Events (AEs) and Serious Adverse Events (SAEs) measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  Safety profile, including SAEs, AEs, deaths, and clinical laboratory abnormalities

OTHER OUTCOMES:
Additional elements of clonal dynamics in CLL | From the start of treatment till end of study, up until the last registered patient has been on pirtobrutinib for 36 months without progressive disease
  Additional genomic profiling and analyses

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No